CLINICAL TRIAL: NCT03205826
Title: Measuring Collateral Ventilation Using Chartis® to Select Patients With Severe Emphysema for Endobronchial Valve Treatment: Conscious Sedation Versus General Anesthesia
Brief Title: Chartis Collateral Ventilation Measurement: Conscious Sedation Versus General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHARTIS sedation
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Emphysema or COPD
Keywords: Emphysema; Bronchoscopic intervention; CHARTIS measurement
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type of sedation used (Other): All patients will undergo two subsequent Chartis measurements. The first measurement will be performed with the patient undergoing conscious sedation and the second measurement with the patient under general anesthesia.
  Interventions: Other: Type of sedation used

INTERVENTIONS:
Other: Type of sedation used — All patients will undergo two subsequent Chartis measurements. The first measurement will be performed with the patient undergoing conscious sedation and the second measurement with the patient under general anesthesia.

SUMMARY:
Rationale: The Chartis® ( Pulmonx, CA, USA) measurement system is a tool to assess interlobar collateral ventilation during bronchoscopy. Assessing collateral ventilation is important when you intend to treat a patient with endobronchial valves. Chartis measurement of collateral ventilation can be performed under both conscious sedation as well as general anesthesia. There is no consensus on what is the preferred method of anesthesia for Chartis measurements in the literature.

Objective: In this project we want to investigate whether there is a difference in Chartis measurement outcomes between these two methods of anesthesia: conscious sedation and general anesthesia.

Study design: This study will be a single center observational study

Study population: The study population exists of patients with severe emphysema who undergo collateral ventilation assessment before bronchoscopic lung volume reduction treatment with one-way endobronchial valves.

Intervention: All patients will undergo two subsequent Chartis measurements. The first measurement will be performed with the patient undergoing conscious sedation and the second measurement with the patient under general anesthesia.

Main study parameters/endpoints: Our primary outcome measure is the failure rate of the Chartis collateral ventilation measurement under general anesthesia versus conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for a bronchoscopic lung volume treatment using one-way valves
* Patient has provided signed informed consent.

Exclusion Criteria:

For safety reasons patients that meet the following criteria will not be included in this study:

1. FEV1 <20%
2. RV/TLC>70%
3. pCO2 >6.5
4. RVSP>40mmHg
5. 6MWT<200m
6. Known intolerance to Lidocaine
7. Any other medical reason/condition that warrants a short procedure (physician judgement )

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Failure rate | Baseline
  The failure rate of the Chartis collateral ventilation measurement under general anesthesia versus conscious sedation.

SECONDARY OUTCOMES:
Chartis measurement duration | Baseline
  To compare the duration of Chartis measurement in patients undergoing conscious sedation versus general anesthesia.
Physician feasibility | Baseline
  To investigate qualitative assessment feasibility for the physician in patients undergoing conscious sedation or general anesthesia.
Influence severity on outcome | Baseline
  To investigate the influence of severity of disease in patients undergoing conscious sedation or general anesthesia.
Influence collateral ventilation status on outcome | Baseline
  To investigate outcome difference in collateral ventilation status in patients undergoing conscious sedation versus general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — d.j.slebos@umcg.nl
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Welling JBA, Klooster K, Hartman JE, Kerstjens HAM, Franz I, Struys MMRF, Absalom AR, Slebos DJ, Barends CRM. Collateral Ventilation Measurement Using Chartis: Procedural Sedation vs General Anesthesia. Chest. 2019 Nov;156(5):984-990. doi: 10.1016/j.chest.2019.07.025. Epub 2019 Aug 15. PMID 31421111